CLINICAL TRIAL: NCT00097747
Title: A Phase 1, Double-blind, Placebo-controlled, Dose Escalation Study of the Safety and Pharmacokinetics of Single Intravenous Doses of Peginesatide in Healthy Volunteers
Brief Title: Safety and Pharmacokinetics of Single Intravenous Doses of Peginesatide in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affymax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AFX01-0401; 2004-001655-11 (EudraCT Number)
Record Dates: First submitted 2004-11-30; First posted 2004-12-01 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Anemia; Chronic Kidney Disease; Chronic Renal Failure; Cancer
Keywords: anemia; chronic kidney disease; CKD; chronic renal failure; CRF; erythropoietin; EPO; erythropoiesis stimulating agent; ESA; Hematide™; hemoglobin; Hb; Hgb; Omontys; peginesatide; red blood cell; red blood cell production
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Failure, Chronic; Neoplasms | interventions — peginesatide; hematide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Single injection administered intravenously
  Interventions: Drug: Placebo
- Peginesatide 0.025 mg/kg (Experimental): Single peginesatide dose of 0.025 milligram per kilogram (mg/kg) administered intravenously.
  Interventions: Drug: peginesatide
- Peginesatide 0.05 mg/kg (Experimental): Single peginesatide dose of 0.05 mg/kg administered intravenously.
  Interventions: Drug: peginesatide
- Peginesatide 0.10 mg/kg (Experimental): Single peginesatide dose of 0.10 mg/kg administered intravenously.
  Interventions: Drug: peginesatide

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: peginesatide
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Peginesatide 0.025 mg/kg; Peginesatide 0.05 mg/kg; Peginesatide 0.10 mg/kg

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics (PK), and minimum pharmacologically active dose of peginesatide in Healthy Volunteers.

DETAILED DESCRIPTION:
This was a Phase 1, double-blind, placebo-controlled trial of peginesatide, an erythropoiesis stimulating agent, with approximately 7 treatment cohorts and 7 healthy volunteer participants per cohort. In each cohort of 7 participants, a ratio of 5:2 participants was randomly assigned to receive a single dose of peginesatide or placebo, respectively, administered as an intravenous infusion. Planned peginesatide dose levels were to escalate by cohort. The study was conducted at a single clinical center.

ELIGIBILITY:
Main eligibility criteria:

* Participant is a healthy male, age ≥ 18 years and ≤ 40 years, with body mass index (BMI) ≥ 18 and ≤ 30 kilograms per squared meter (kg/m^2), and weight ≥ 50 and ≤ 95 kilograms (kg)
* Participant has hemoglobin of ≤ 16 grams per deciliter (g/dL) at the time of study entry
* Participant has normal iron stores

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2004-08; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | 28 Days

SECONDARY OUTCOMES:
PK parameters | 28 Days
Pharmacodynamic (PD) parameters | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Affymax, Study Director — Affymax, Inc.
Locations (1):
- Research Facility, London, United Kingdom